CLINICAL TRIAL: NCT05149326
Title: A Multicenter, Randomized, Double-Blind Phase III Study to Assess the Efficacy and Safety of KN046 Combined With Gemcitabine and Nab-Paclitaxel Versus Placebo Combined With Gemcitabine and Nab-Paclitaxel in First Line Advanced Pancreatic Ductal Adenocarcinoma Subjects (ENREACH-PDAC-01).
Brief Title: KN046 in Subjects With Advanced Pancreatic Ductal Adenocarcinoma.
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Alphamab Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KN046-303
Record Dates: First submitted 2021-11-26; First posted 2021-12-08 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Advanced Pancreatic Ductal Adenocarcinoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental)
  Interventions: Drug: KN046
- Control arm (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: KN046 — KN046+Nab-Paclitaxel+Gemcitabine In combine therapy stage, KN046 is 5 milligram per kilogram, every 2 weeks. In maintain stage, KN046 is 5 milligram per kilogram, every 2 weeks.
  Arms: Experimental arm
Drug: placebo — placebo+Nab-Paclitaxel+Gemcitabine In combine therapy stage, placebo is 5 milligram per kilogram, every 2 weeks. In maintain stage, placebo is 5 milligram per kilogram, every 2 weeks.
  Arms: Control arm

SUMMARY:
This study is a multicenter, randomized, double-Blind Phase III Study to compare the clinical efficacy and safety of KN046 plus gemcitabine and nab-paclitaxel versus placebo plus gemcitabine and nab-paclitaxel in subjects with advanced pancreatic ductal adenocarcinoma who have not previously received systemic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18, male or female;
* Has histologically or cytologically confirmed pancreatic ductal adenocarcinoma (PDAC);
* Has not received prior systemic treatment for their locally advanced or metastatic PDAC;
* Has presence of measurable disease as defined by Response Evaluation Criteria in Solid Tumours (RECIST 1.1);
* Has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Status;
* Has a life expectancy of at least 3 months;
* Has adequate organ function;
* If female of childbearing potential, have a negative serum pregnancy test within 7 days prior to first trial treatment;
* If female of childbearing potential or a male subject with a partner with childbearing potential, be willing to use a highly effective method of contraception (with a failure rate of less than 1.0% per year) from first study treatment to 24 weeks after completion of the trial treatment.

Exclusion Criteria:

* Untreated active CNS metastasis or leptomeningeal metastasis.
* Is currently participating and receiving an investigational drug or has participated in a study of an investigational drug within 4 weeks or within 5 times of half-life (no less than 2 weeks), whichever is shorter prior to the first dose of trial treatment;
* Has received other anti-tumor treatment within 4 weeks or within 5 times of half-life (no less than 2 weeks), whichever is shorter prior to the first trial treatment;
* Major surgery for any reason, except diagnostic biopsy, within 4 weeks of the first administration of trial treatment and/or if the subject has not fully recovered from the surgery within 4 weeks of the first administration of trial treatment;
* Curative radiation within 3 months of the first dose of trial treatment. Radiation to more than 30% of the bone marrow or with a wide field of radiation should not be used within 4 weeks prior to the first administration of trial treatment;
* Subjects receiving immunosuppressive agents (such as steroids) for any reason should be tapered off these drugs before initiation of trial treatment (with the exception of subjects with adrenal insufficiency, who may continue corticosteroids at physiologic replacement doses, equivalent to < 10 mg prednisone daily, inhaled steroids and topical use of steroids);
* Vaccination within 28 days of the first administration of trial treatment, except for administration of inactivated vaccines (e.g., inactivated influenza vaccines);
* Has interstitial lung disease, or a history of pneumonitis that required oral or intravenous glucocorticoids to assist with management;
* History or current active autoimmune disease that might deteriorate when receiving an immunostimulatory agent；
* Previous malignant disease History of uncontrolled intercurrent illness Prior therapy with any antibody/drug targeting T cell coregulatory proteins Known severe hypersensitivity reactions to antibody drug；
* Is pregnant or breastfeeding;
* Other medical conditions that at the discretion of investigator interfere with the requirements of the trial in terms of safety or efficacy evaluation, or treatment compliance.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Estimated)
Dates: Start 2022-01-20 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | up to 2 years
  OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the interim analysis were censored at the date of the last follow-up.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | up to 2 years
  Time between randomization to date of disease progression or death due to any cause.
Overall response rate (ORR) | up to 2 years
  Complete Response or Partial Response according to RECIST

CONTACTS AND LOCATIONS:
Locations (65):
- China (65):
  - The Second Hospital Of Anhui medical University, Hefei, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The Southwest Hospital of AMU, Chongqing, Chongqing Municipality
  - The Third Affiliated Hospital of Army Medical University, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital,Sun Yat-sen University, Guangzhou, Guangdong
  - Affiliated Cancer Hospital of Guangxi Medical University, Nanning, Guangxi
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Union Hospital Tongji Medical College Huazhong University of Science And Technology, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - The Affiliated Hospital Of XuZhou Medical University, Xuzhou, Jiangsu
  - First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Shandong Cancer Hospital, Jinan, Shandong
  - Shandong Provincial Hospital, Jinan, Shandong
  - Affiliated Hospital of Jining Medical University, Jining, Shandong
  - LINYI Cancer Hospital, Linyi, Shandong
  - Linyi City People Hospital, Linyi, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Weifang People'S Hospital, Weifang, Shandong
  - Shanghai Changhai Hospital, Shanghai, Shanghai Municipality
  - Yueyang Hospital of Integrated Traditional Chinese and Western Medicine , Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Shanxi Cancer hospital, Taiyuan, Shanxi
  - Shanxi Provincial People's Hospital, Taiyuan, Shanxi
  - the First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hosipital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Zhejiang Provincial People's hospital, Hangzhou, Zhejiang
  - Jiaxing Second Hospital, Jiaxing, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No